CLINICAL TRIAL: NCT02474732
Title: Assessment of User Comprehension of the BeActive™Brace User Guide
Brief Title: Usability Study for the Beactive Brace Instructions for Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benjamin L. England and Associates, LLC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: C15-0419
Record Dates: First submitted 2015-06-12; First posted 2015-06-18 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Lower Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Braces

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Usability (Other): Determine if the subjects are able to understand and follow the directions to apply the Beactive Brace.
  Interventions: Device: Beactive(r) Brace

INTERVENTIONS:
Device: Beactive(r) Brace — Determine if the subjects are able to understand and follow the directions to apply the Beactive Brace.

SUMMARY:
FDA requires that the user's guide be provided with any over-the-counter (OTC) medical device. It is beneficial to demonstrate that the user's guide for a new medical device is broadly comprehensible where the device will be provided without prescription and direct physician counseling. Therefore, a population of subjects will be tested to determine whether they can properly use the BeActive Brace device after reading the user's guide.

DETAILED DESCRIPTION:
The primary objective of this clinical trial is to evaluate the ability of approximately 40 literate adults to understand the label instructions for deploying the Beactive(r) Brace device as described in the user's guide, without physician direction. The primary endpoint of this clinical trial is the successful completion of all essential tasks required for Beactive(r) Brace deployment by a subject.

Subjects will be seated at a table facing a video camera, so Investigators and the Sponsor may observe the subject via closed circuit television. Subjects will be given the user's guide for the Beactive(r) Brace device. The subject will then be asked to deploy the Beactive(r) Brace device according to their understanding following the user's guide. For this clinical trial, deploying is defined as completing the following two tasks.

1. Applying the Beactive(r) Brace device to the knee area according to the user's guide.
2. Correctly positioning the pressure pad according to the user's guide.

If the tasks can be completed with no intervention, the subject would be judged to have a "comprehensive" level of success. If intervention was required and helpful, and the subject was able to complete all essential tasks, the level of success would be judged "sufficient." The steps where intervention took place will be recorded.

Intervention will be allowed and documented if subjects have difficulty with a specific task. The subject will raise their hand and a technician will be available for assistance. The frequency and type of intervention will be documented.

A Study Coordinator will complete an observer questionnaire for each subject based on their observation of each subject's ability to use the Beactive device correctly. Each subject will complete a user questionnaire, which will confirm their understanding of the user's guide and give them the opportunity to provide feedback and suggestions for improving the user's guide.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be male or female, between the ages of ages 22 to 79 years (inclusive);
* Subjects must understand and execute an Individual Consent Form (ICF) and complete a Medical History Form;
* Subjects must be in general good health, except for back pain;
* Subjects must have a history of lower back pain with radiating pain down the leg;
* Subjects must have completed the 10th grade and must be able to read and comprehend English;
* Subjects must be willing to report any medications taken during the trial and refrain from taking medication that might reduce back pain; and
* Subjects must be considered reliable and capable of following directions.

Exclusion Criteria:

* Subjects in ill health or taking medication, other than birth control, which could influence the purpose,integrity or outcome of the trial; or
* Subjects having any visible skin disease, which might be confused with a skin reaction from the test material.

Ages: 22 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-02; Primary Completion 2015-02 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Number of Subjects Correctly Following Instructions for Use | Five minutes
  Subjects were observed as they read the instructions for use and applied the Beactive(r) Brace.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Caswell, Study Director — Consumer Product Testing Compahy, Inc.

IPD SHARING:
Plan to Share IPD: No
Redacted individual participant data is available through the Freedom of Information Act process through the FDA